CLINICAL TRIAL: NCT05833984
Title: A Phase 1b/2 Dose Escalation and Expansion Study Evaluating the Safety, Tolerability, and Efficacy of IMM01 Plus Tislelizumab in Patients With Advanced Solid Tumors and Lymphomas
Brief Title: Safety and Efficacy of IMM01 Plus Tislelizumab in Patients With Advanced Solid Tumors and Lymphomas
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMM01-04
Record Dates: First submitted 2023-03-27; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Solid Tumor; Classic Hodgkin Lymphoma
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Dose Escalation Part (Experimental): Mutiple dose level cohorts in the dose escalation part
  Interventions: Drug: IMM01; Drug: Tislelizumab
- Head and neck squamous cell carcinoma, nasopharyngeal carcinoma (Experimental): Dose expansion cohort with IMM01 plus Tislelizumab
  Interventions: Drug: IMM01; Drug: Tislelizumab
- Ovarian carcinoma (Experimental): Dose expansion cohort with IMM01 plus Tislelizumab
  Interventions: Drug: IMM01; Drug: Tislelizumab
- Non small cell lung carcinoma, small cell lung carcinoma (Experimental): Dose expansion cohort with IMM01 plus Tislelizumab
  Interventions: Drug: IMM01; Drug: Tislelizumab
- Hepatocellular carcinoma (Experimental): Dose expansion cohort with IMM01 plus Tislelizumab
  Interventions: Drug: IMM01; Drug: Tislelizumab
- Other solid tumors (Experimental): Dose expansion cohort with IMM01 plus Tislelizumab
  Interventions: Drug: IMM01; Drug: Tislelizumab
- Classic hodgkin lymphoma (Experimental): Dose expansion cohort with IMM01 plus Tislelizumab
  Interventions: Drug: IMM01; Drug: Tislelizumab

INTERVENTIONS:
Drug: IMM01 — IMM01 (1.0, 1.5, 2.0 mg/kg) QW IV in the dose escalation part. IMM01 (dose determined in the dose escalation part) QW IV in the dose expansion part.
  Other Names: SIRPα Fc
Drug: Tislelizumab — Tislelizumab 200mg Q3W IV

SUMMARY:
This is an open-label, multicenter, phase 1b/2 trial of IMM01 (SIRPα Fc) plus tislelizumab in patients with advanced solid tumors and lymphomas.

DETAILED DESCRIPTION:
This open-label, multicenter, phase 1b/2 trial is conducted to evaluate the safety, tolerability and preliminary activity in patients with advanced solid tumors and lymphomas. This trial includes two parts: the phase 1b dose escalation part and the phase 2 dose expansion part.

In the dose escalation part with a standard 3+3 design, IMM01 (1.0, 1.5, 2.0 mg/kg) was administered once a week and tislelizumab (200mg) was administered once every 3 weeks.

In the dose expansion part, IMM01 (the dose determined in the dose escalation part) was administered once a week and tislelizumab (200mg) was administered once every 3 weeks. And the cohorts includes HNSCC, NSCLC, SCLC, R/R cHL and others.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female
2. Life expectancy≥12 weeks;
3. Phase 1b: Patients with advanced solid tumors diagnosed by histology or cytology, who have been failure to previous standard treatments; Phase 2: Patients with HNSCC, NPC, OC, NSCLC, SCLC, HCC, cHL and other solid tumors diagnosed by histology or cytology, who have been failure to first-line standard treatment (including PD-1/L1) at least;
4. ECOG PS of 0 or 1;
5. Adequate organs function, including bone marrow, hepatic, renal, cardiac, coagulation.
6. Adverse events associated with previous anti-tumor therapy have returned to≤ grade 1(NCI CTCAE V5.0);

Exclusion Criteria:

1. Previous treatment with CD47 inhibitor/SIRPαinhibitor or fusion protein;
2. Patients with symptomatic or progressive central nervous system (CNS) metastasis;
3. Uncontrolled hypertension, pulmonary hypertension or unstable angina, myocardial infarction within 6 months prior to administration; a history of chronic heart failure (NYHA G3/4); severe arrhythmia;
4. A history of arterial thrombosis, deep venous thrombosis and pulmonary embolism within 3 months prior to administration;
5. A history of moderate or severe dyspnea, interstitial lung disease (ILD) or servre pneumonia, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency;
6. With other malignant tumors;
7. Diseases that may cause gastrointestinal bleeding or perforation;
8. Uncontrollable pleural, peritoneal or pericardial effusions;
9. A history of immunodeficiency;
10. A history of autoimmune diseases;
11. Uncontrolled severe active infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2024-02-07 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity in dose escalation part | DLT observation 21 days
MTD/RP2D in dose escalation part | DLT observation 21 days
ORR in dose expansion part | up to 12 months

SECONDARY OUTCOMES:
TRAEs | up to 12 months
PFS | up to 12 months
DOR | up to 12 months
DCR | up to 12 months
Cmax | up to 12 months
T1/2 | up to 12 months
AUC | up to 12 months
ADA | up to 12 months

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Zhejiang Cancer Hospital, Hangzhou
  - Shandong Provincial Institute of Cancer Prevention and Treatment, Jinan
  - The Third Affiliated Hospital of Qiqihar Medical University, Qiqihar
  - Shanghai Chest Hospital, Shanghai
  - Henan Cancer Hospital, Zhengzhou